CLINICAL TRIAL: NCT07177040
Title: Effect of SNAG Versus Maitland Techniques in the Management of Non-Specific Low Back Pain
Brief Title: Effect of Two Different Mobilization Techniques in the Treatment of Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ehab Mohamed Kamel Ahmed (Other)
Collaborators: The Scientific Research Deanship, University of Ha'il (Unknown)
Responsible Party: Sponsor-Investigator, Ehab Mohamed Kamel Ahmed, Department of Public Health, College of Public Health and Health Informatics, University of Hail, Ha'il, Saudi Arabia, University of Hail
Organization: University of Hail (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2025-858
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Non-specific Low Back Pain (NSLBP)

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland (Active Comparator): Participants will receive Maitland technique therapy
  Interventions: Procedure: Maitland; Procedure: SNAG
- SNAG (Active Comparator): Participants will receive SNAG therapy based on the Mulligan Concept
  Interventions: Procedure: Maitland; Procedure: SNAG

INTERVENTIONS:
Procedure: Maitland — Maitland technique therapy, which consists of passive mobilizations applied to the lumbar facet joints in an anterocranial direction while the patient is in a prone lying position
Procedure: SNAG — The technique involves applying a sustained glide to the lumbar facet joints while the patient is in a sitting position, and the pelvic girdle will be stabilized by a belt. Then the therapist will ask the patient for active forward flexion of the spine while the pressure on the facet joint is maintained during the movement till its end
  Other Names: sustained natural apophyseal glide

SUMMARY:
Non-specific low back pain (NSLBP) is extensively musculoskeletal conditions, where manual therapy techniques have been widely employed in its management, but their short term efficacy in chronic low back pain still need more investigations. Objective: This study aimed to discuss the SNAG versus Maitland techniques in the management of NSLBP. Methods: 60 patients with chronic NSLBP will share in the study. Sessions will be conducted 3 times per week for 4 weeks. The outcomes will be evaluated for pain by the numerical rating pain scale (NPRS), disability through Oswestry Disability Index, flexion range of motion by back range of motion device, postural stability by Biodex system will be assessed at baseline, immediately post-intervention, and at a four-week follow-up

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 40 years.
* Diagnosed with chronic NSLBP persisting for more than three months.
* Pain intensity between 3 to 6 on the Visual Analog Scale (VAS) during lumbar extension in a sitting position.
* Oswestry Disability Index (ODI) score between 20% to 40%.
* Restriction of the movement only in flexion ROM with the ability to perform at least 40° of trunk flexion.

Exclusion Criteria:

* Specific causes of low back pain (e.g., herniated disc, spinal stenosis).
* History of spinal surgery or trauma.
* Neurological deficits or systemic diseases affecting the musculoskeletal system.
* Pregnancy.
* Current participation in other physiotherapy programs.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  The NPRS will be used to evaluate the level of pain by selecting a number on a rating scale, ranging from 0 (no pain) to 10 (worst and unbearable pain).

SECONDARY OUTCOMES:
Functional disability | 4 weeks
  Assessed by the Oswestry Disability Index (ODI) where according to the scale the disability will be indicated as follow: 0-4 no disability, 5-14 mild disability, 5-24 moderate disability, 25-34 severe disability, and 35-50 complete disability
Lumbar flexion range of motion | 4 weeks
  Measured using a Back range of motion (BROM)
overall stability index (OSI) | 4 weeks
  Repositioning error evaluated through proprioceptive testing provided by the Biodex Balance System, no need for cut off) as the measurement differences will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Clinics, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
All the data will be obtained from the experiment is under the protection of the Scientific Research Deanship, University of Ha'il, Saudi Arabia as this project is funded from it with number RG-20 202.